CLINICAL TRIAL: NCT06399926
Title: A Open-label, Random, Multi-central Prospective Cohort of Observation Study on the Efficacy and Safety of Intraventricule Pemetrexed Disodium Via Ommaya Reservoir
Brief Title: Efficacy and Safety of Intraventricule Pemetrexed Disodium Administered Via Ommaya Reservoir
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: First People's Hospital of Chenzhou (Other); Xiangtan Central Hospital (Other)
Responsible Party: Principal Investigator, Bin Li, MD, Associated professor, Xiangya Hospital of Central South University
Other Study IDs: 2023121058
Record Dates: First submitted 2024-03-18; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Leptomeningeal Metastasis; Lung Cancer
Keywords: Leptomeningeal Metastasis; Ommaya reservoir; Pemetrexed
MeSH Terms: conditions — Meningeal Carcinomatosis; Lung Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid(CSF) supernatants are retained for the detection of cytokines and Pemetrexed concentration.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pemetrexed 20mg: Pemetrexed 20mg every 24 hours for 72 hours every 2 weeks until efficacy evaluated remission or stable ; change to every 3 weeks.
  Interventions: Drug: Pemetrexed injection; Drug: Pemetrexed
- Pemetrexed 30mg: Pemetrexed 30mg D1 every week until efficacy evaluated remission or stable ; change to every 3 weeks.
  Interventions: Drug: Pemetrexed injection; Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed injection — Group 1（20mg）:induction stage is 20 mg per 24 hours for 72 hours, every 2 weeks; consolidation stage is 20mg per 24 hours for 72 hours, every 3 weeks.
  Other Names: Alimta
Drug: Pemetrexed — Group 2（30mg）:induction stage is 30 mg D1，every week.Consolidation stage is 30 mg D1,every 3 weeks.
  Other Names: Alimta

SUMMARY:
This is a open-label, multi-center prospective observation study for the efficacy and safety of intraventricle pemetrexed disodium via ommaya reservoir in the treatment of leptomeningeal metastasis with lung cancer who have failed at least one targeted therapy. In detail: At least the treatment failure was after third-generation EGFR-TKIs in EGFR-mutated lung cancer; or at least the treatment failure was after second-generation ALK-TKIs in ALK-mutated lung cancer; or at least the treatment failure was after one-line of targeted-TKIs in ROS1-mutated non-squamous non-small lung cancer.

DETAILED DESCRIPTION:
Participants were randomizedly assigned in cohort 1 who will be given pemetrexed 20mg every 24 hours for 72 hours every 2 weeks,or in cohort 2 will be given pemetrexed 30mg once a week.

It was designed for two stages on treatment course. Induction therapy: Efficacy evaluation every 2 cycles, and confirm the efficacy at the next cycle. If at the next cycle, the efficacy result changed (such as SD or PR after initial PD; or PD after initial SD or PR; the second time of efficacy assess was required）. If the CSF cytology at the time of the efficacy evaluation was negative, one more cycle was required to confirm the CSF cytology.

Consolidation: If the efficacy is remission(including complete remission, obvious remission, or partial remission) or stable disease for initial timepoint and the timepoint of the confirmed evaluation; then the patient will be advanced to the stage of consolidation treatment. Participants in cohort 1 who will be given pemetrexed 20mg every 24 hours for 72 hours every 3 weeks. Participants in cohort 2 will be given pemetrexed 30mg every 3 weeks. Until the toxicity is intolerable, or disease progression.

Cross over： Compared the first 4 enrolled cases in each group; the comprehensive evaluation(including efficacy, cytology negative, toxicity) in better group(50% higher efficacy or 50% less toxicity) will be the following cohort, to which the other one will crossover.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed pathologic diagnosis (histologic type of non-squamous non-small cell lung cancer in the primary lesion or metastatic lesion) with definitely genetic testing results (EGFR/ALK/ROS1);
2. In accordance with the CSCO Guidelines for the Diagnosis and Management of Central Nervous System Tumors, and the EANO-ESMO diagnostic criteria: a diagnosis of type I meningeal metastatic carcinoma is made when cerebrospinal fluid cytology testing reveals anisocytosis (3 consecutive tests are required if the cerebrospinal fluid cytology testing is initially negative for the patient) (one study showed that the specificity of anisocytosis in diagnosing meningeal metastases in patients with solid tumors was 100%) or meningeal lesions Biopsy confirms the diagnosis. (Type IIA-C meningeal metastases: negative or atypical cerebrospinal fluid cytology, MRI showing linear or/and nodular meningeal enhancement^ with typical clinical symptoms*).

   * MRI: at least 1.5T; demonstrates sulcal, smear, or linear ventricular enhancement, cranial nerve root enhancement or nodular meningeal enhancement, or cauda equina spinal enhancement; control enhancement T1-weighted sequences and Flair sequences; nodularity is defined as foci of ≥ 5x10mm enhancement; sequences of choice: cranial planar enhancement + T2Flair (enhancement) or and total spinal planar enhancement (when suspicion of spinal involvement); 3D T1 enhancement (involved cranial nerves - optional); cerebrospinal fluid flow imaging (functional or anatomic).

     * Typical clinical manifestations: headache, nausea, vomiting; epilepsy; mental changes, gait difficulties; cranial nerve damage (diplopia, visual abnormalities, hearing abnormalities, facial nerve palsy, difficulty chewing, difficulty swallowing, choking, etc.); neurogenic signs (cauda equina symptoms, mainly perineal numbness, tingling, defecation and urination disturbances, weakness or incomplete paralysis of both lower limbs); sensorimotor defects of the limbs; cervical back Radicular pain; be careful to differentiate from signs and symptoms of brain parenchymal metastases, extracranial disease, treatment-related adverse effects, and non-tumor comorbidities.

       3. Based on the guideline-driven first-line choice of TKI agents for gene-positive patients, enrolment would therefore require: failure of at least three generations of EGFR-TKIs for patients with EGFR mutations; failure of at least second-generation ALK inhibitors for ALK mutations; and failure of at least one ROS1 inhibitor for ROS1 mutations.

       4. No contraindication to Ommaya capsule implantation. 5. Female subjects who are capable of becoming pregnant must agree to use reliable contraception throughout the trial; male subjects whose female partner is capable of becoming pregnant must agree to use reliable contraception throughout the trial.

       6. patients must sign an informed consent form and must be willing and able to comply with visits, treatment regimens, laboratory tests and other requirements as specified in the study protocol

Exclusion Criteria:

1. HBsAg-positive patients may be enrolled, but patients with higher than normal viral copy number or HBcAb-positive patients should receive effective anti-HBV treatment until 6 months after the end of the trial. HCV RNA carriers may be enrolled, but need to receive effective anti-HCV treatment throughout the trial, and continue to receive effective anti-HCV treatment until 6 months after the end of the trial.
2. human immunodeficiency virus (HIV) infection.
3. significant extracranial lesion progression or extensive extracranial lesions causing severe symptoms that cannot be effectively treated.
4. patients with extreme emaciation or cachexia.
5. Extensive parenchymal brain lesions with severe symptoms that cannot be effectively treated.
6. patients with other malignant tumors that are currently undergoing treatment.
7. have received or will receive a live vaccine within 30 days prior to signing the informed consent form.
8. other conditions that, in the judgment of the investigator, may affect subject safety or trial compliance, including symptomatic heart failure, unstable angina, myocardial infarction, active infections (including tuberculosis infections) requiring systemic therapy; or severe organ dysfunction, with creatinine clearance <45 ml/min calculated from glomerular filtration rate by the Cockcroft-Gault formula or by the Tc99m-DPTA serum clearance method; an absolute neutrophil count <0.5 x 109/L; a platelet count <25 x 109/L, or in patients with severe active visceral bleeding; or severe Abnormal liver function (bilirubin greater than 3.0 times upper limit of normal; AST and ALT greater than 5.0 times upper limit of normal).
9. patients with known hypersensitivity to pemetrexed with a history of serious adverse reactions, and patients with potentially life-threatening conditions for reuse.
10. pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-squamous non-small cell lung cancer with oncogene-driven and failed at least one-line of targeted therepy ( EGFR/ALK/ROS1); At least failure after third-generation EGFR-TKIs in EGFR-mutated lung cancer. At least failure after second-generation ALK-TKIs in ALK-mutated lung cancer. At least failure after one line of targeted-TKIs in ROS1-mutated non-squamous non-small lung cancer.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate，ORR | 3 months
  ORR is the ratio of the patients who achieve the complete remission(CR), obvious remission(OR), or partial remission(PR) to the included patients eligible for efficacy assessment. complete remission(one of the following items): normal RANO；normal Glasgow Coma Scale；KPS≥90.
  obvious remission(one of the following items): the improvement of at least 70% items on the RNAO examinations; Glasgow Coma Scale≥12 or at lease 3 scores increase compared to baseline; KPS≥70 or at lease 30 scores increase compared to baseline.
  partial remission(one of the following items)：the improvement of at least 50% items on the RNAO examinations; Glasgow Coma Scale≥9 or at lease 2 scores increase compared to baseline; KPS 50-70 or at lease 20 scores increase compared to baseline.

SECONDARY OUTCOMES:
Disease control rate,DCR | 2 years
  DCR is the ratio of the patients who achieve the CR, OR, PR,or SD to the included patients eligible for efficacy assessment. complete remission(one of the following items): normal RANO；normal Glasgow Coma Scale；KPS≥90.
  obvious remission(one of the following items): the improvement of at least 70% items on the RNAO examinations; Glasgow Coma Scale≥12 or at lease 3 scores increase compared to baseline; KPS≥70 or at lease 30 scores increase compared to baseline.
  partial remission(one of the following items)：the improvement of at least 50% items on the RNAO examinations; Glasgow Coma Scale≥9 or at lease 2 scores increase compared to baseline; KPS 50-70 or at lease 20 scores increase compared to baseline.
  stable disease (one of the following items ):the improved items on the RNAO examinations less than 50%; the change of Glasgow Coma Scale within 1 score compared to baseline; the change of KPS within 10 scores.
progression-free survival，PFS | 2 years
  time to the progression of disease. Progression of disease(one of the following items): The deterioration of at least 25% items on the RNAO examinations; the drop of Glasgow Coma Scale more than 1 score compared to baseline; the drop of KPS score more than 10 scores.
overall survival,OS | 2 years
  time to the death or loss of follow-up
CSF cytology clearance | 2 years
  negative results using glass slide centrifugation accompanied with staining
Adverse effect（AE） and severe Adverse effect(SAE) | 2 years
  number of participants with treatment-related adverse events or severe adverse effect as assessed by CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: bin Li, doctor, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided
we will share the some dates to the website:http://www.medresman.org.cn/login.aspx or publication of results of clinical trials in the form of papers

REFERENCES:
- [Result] Maynard A, McCoach CE, Rotow JK, Harris L, Haderk F, Kerr DL, Yu EA, Schenk EL, Tan W, Zee A, Tan M, Gui P, Lea T, Wu W, Urisman A, Jones K, Sit R, Kolli PK, Seeley E, Gesthalter Y, Le DD, Yamauchi KA, Naeger DM, Bandyopadhyay S, Shah K, Cech L, Thomas NJ, Gupta A, Gonzalez M, Do H, Tan L, Bacaltos B, Gomez-Sjoberg R, Gubens M, Jahan T, Kratz JR, Jablons D, Neff N, Doebele RC, Weissman J, Blakely CM, Darmanis S, Bivona TG. Therapy-Induced Evolution of Human Lung Cancer Revealed by Single-Cell RNA Sequencing. Cell. 2020 Sep 3;182(5):1232-1251.e22. doi: 10.1016/j.cell.2020.07.017. Epub 2020 Aug 20. PMID 32822576
- [Result] Thakkar JP, Kumthekar P, Dixit KS, Stupp R, Lukas RV. Leptomeningeal metastasis from solid tumors. J Neurol Sci. 2020 Apr 15;411:116706. doi: 10.1016/j.jns.2020.116706. Epub 2020 Jan 23. PMID 32007755
- [Result] Mack F, Baumert BG, Schafer N, Hattingen E, Scheffler B, Herrlinger U, Glas M. Therapy of leptomeningeal metastasis in solid tumors. Cancer Treat Rev. 2016 Feb;43:83-91. doi: 10.1016/j.ctrv.2015.12.004. Epub 2015 Dec 24. PMID 26827696
- [Result] Ommaya AK. Subcutaneous reservoir and pump for sterile access to ventricular cerebrospinal fluid. Lancet. 1963 Nov 9;2(7315):983-4. doi: 10.1016/s0140-6736(63)90681-0. No abstract available. PMID 14059058
- [Result] Montes de Oca Delgado M, Cacho Diaz B, Santos Zambrano J, Guerrero Juarez V, Lopez Martinez MS, Castro Martinez E, Avendano Mendez-Padilla J, Mejia Perez S, Reyes Moreno I, Gutierrez Aceves A, Gonzalez Aguilar A. The Comparative Treatment of Intraventricular Chemotherapy by Ommaya Reservoir vs. Lumbar Puncture in Patients With Leptomeningeal Carcinomatosis. Front Oncol. 2018 Nov 20;8:509. doi: 10.3389/fonc.2018.00509. eCollection 2018. PMID 30524956